CLINICAL TRIAL: NCT05912166
Title: Meditation, Education, Navigation, & Training Using eHealth: Cancer Adaptation Through Learning Mindful Awareness
Acronym: MenteCalma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Victorson, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NU 23CC02; 3R01CA262357-02S1 (NIH)
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Cancer
Keywords: cancer; young adult; e-health; mindfulness; remote-delivered; Spanish-language; international; Colombia
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The researchers will collect implementation feasibility and acceptability data of the 9-week Spanish-language Wakeful app in a mixed sample of young adult cancer survivors (n=30) between 18-39, using a single arm pre-post test design. Following consent, participants will be immediately directed to a secure Redcap assessment URL to complete the T1 assessment. Next, participants will be sent an email to access the Wakeful web app where they will watch a brief video orientation and begin the 9-week self-directed course. After 9 weeks, participants will be emailed a secure URL to complete the T2 assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wakeful Spanish (Experimental): Wakeful Spanish is the Spanish-language version of Wakeful, developed at Northwestern University. It is a self-directed 9-week digital mindfulness course closely aligned with traditional 8-week Mindfulness-based Stress Reduction (MBSR) programs.
  Interventions: Behavioral: Wakeful Spanish

INTERVENTIONS:
Behavioral: Wakeful Spanish — Wakeful Spanish is the Spanish-language version of Wakeful, a self-directed 9-week digital mindfulness course closely aligned with traditional 8-week Mindfulness-based Stress Reduction (MBSR) programs. Wakeful makes one new class available to users each week for 9 weeks. Users receive weekly email notifications from Wakeful informing them when a new class is available. Estimated class duration is 1-1.5 hours.
  With Wakeful, users can -
  1. Write what they observed during meditations.
  2. Be guided by videos/audios through breathing exercises and gentle stretching.
  3. See what others experienced and their tips for overcoming challenges.
  4. Access videos/audios that explain how mindfulness benefits the body and mind.
  5. Receive suggestions on meditations to do during the week
  6. Set an intention for the week based on class content.

SUMMARY:
The purpose of this international oncology research includes the following three aims:

* Aim 1. Expand and strengthen the existing research partnership with investigators from Centro Javeriano de Oncología, Pontificia Universidad Javeriana, and Hospital Universitario San Ignacio in Bogotá, Colombia.
* Aim 2. Evaluate the implementation feasibility and acceptability of the 9-week Spanish-translated mindfulness app, Wakeful, in a mixed Colombian young adult cancer patient sample.
* Aim 3. Translate and record professional Spanish-language voice overs for all new STU00210628 content for future implementation.

DETAILED DESCRIPTION:
The purpose of this international oncology research includes the following three aims:

* Aim 1. Expand and strengthen the existing research partnership with investigators from Centro Javeriano de Oncología, Pontificia Universidad Javeriana, and Hospital Universitario San Ignacio in Bogotá, Colombia.
* Aim 2. Evaluate the implementation feasibility and acceptability of the 9-week Spanish-translated mindfulness app, Wakeful, in a mixed Colombian young adult cancer patient sample.
* Aim 3. Translate and record professional Spanish-language voice overs for all new STU00210628 content for future implementation.

The research is a collaborative study. All research activities, except implementation of the Wakeful intervention-related research activities, will be conducted by Centro Javeriano de Oncologia research staff, and data collection will take place online via Zoom and REDCap accounts. Northwestern research staff will be involved in Wakeful app intervention related activities (i.e., conducting the Wakeful orientation via Zoom; providing Wakeful intervention management and technical support; data collection via the Wakeful app; sending reminders via the Wakeful app, following-up with participants who have not used the Wakeul app in 14 days; and data analysis). The following are the study sites: Northwestern University and Centro Javeriano de Oncologia. This study will not seek sIRB or reliance agreement. Each site will seek local IRB approval.

The research investigators will conduct a pre-post feasibility study. Thirty men and women will complete a 9-week online course. Participants will be assessed at baseline just prior to the start of the course (T1), followed by assessments at 9 weeks (T2). Following consent, participants will be immediately directed to a secure REDCap survey URL to complete the T1 (baseline) survey. The survey will take approximately 20-30 minutes to complete. Next, participants will receive an email invitation to participate in a Wakeful orientation via Zoom, during which they will receive an email from the Wakeful app inviting them to register. By clicking the "Create Password" button in the email invitation, they will be directed to the Wakeful registration page where they will create a unique username and password. Wakeful will then prompt them to confirm their username and password and sign in. Once they sign in, Wakeful will prompt them to watch a brief video orientation and begin the 9-week self-directed course. Within 24 hours of completing the 9 Wakeful classes, a participant will receive an email with instructions and a link to complete the T2 survey. At the end of participation, no other information will be collected by the app; however, participants will still have access to specific features of the app (i.e., the mindfulness videos for review and the timer for continued practice) in the event they would like to continue their mindfulness practice after study participation.

Spanish-language assessments will occur over the internet through a secure REDCap platform. Outcome measures include: socio-demographic and clinical information (gathered at T1); feasibility metrics (gathered on an ongoing basis throughout the study); acceptability and satisfaction metrics (gathered at T2); usability metrics (gathered on an ongoing basis throughout the study); and health related quality of life and wellbeing measures (gathered at all time-points unless otherwise indicated).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer
* Age 18-39 years at time of enrollment
* Under treatment or within 3 years of having completed primary cancer treatment (i.e., surgery, chemotherapy, or radiation) at time of enrollment
* Access to a device with Wifi (e.g., smartphone, computer, tablet)
* Fluency in spoken and written Spanish

Exclusion Criteria:

* Bedridden, or physical debilitation such that study participation would not be feasible or would create undue hardship
* Inability to provide informed consent
* Prisoners or other detained individuals at time of enrollment

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2024-09-29 (Actual)

PRIMARY OUTCOMES:
Implementation feasibility measured by enrollment rate | continuously for 9 weeks
  This indicator of implementation feasibility for the intervention delivered is defined by the overall enrollment rate being >/= 70% (e.g., total number of individuals enrolled/total number approached). Enrollment rate will be tracked continuously during the 9-week study.
Implementation feasibility measured by retention rate | continuously for 9 weeks
  This indicator of implementation feasibility for the intervention delivered is defined by the retention rate being >/= 70% (e.g., total number of participants who drop out/ total number enrolled). Retention rate will be tracked continuously during the 9-week study.
Implementation feasibility measured by completion rate | continuously for 9 weeks
  This indicator of implementation feasibility for the intervention delivered is defined by the overall completion rate being >/= 70% (e.g., total number of individuals completed/total number enrolled). Completion rate will be tracked continuously during the 9-week study.
Acceptability of the Wakeful program as measured by a post-intervention evaluation survey | post-intervention
  Acceptability will be measured using a Likert-type survey assessing participant enjoyment, satisfaction, perceived benefit, and ease of use. Acceptability is defined as >/= 70% of survey responses in affirmation of this.
Acceptability of the Wakeful program as measured by mindfulness reflections | continuously for 9 weeks
  Acceptability of the Wakeful program as measured by mindfulness reflections written by participants in the Wakeful app will be collected continuously during the 9-week study. Written mindfulness reflections downloaded, de-identified, and coded using Dedoose, a collaborative, web-based application that facilitates all types of research data management and analysis. The study team will identify common themes, create definitions, and develop coding rules regarding specific group comments. The comments will then be compiled and summarized in frequency tables denoting the number of times responses were made. Results will be summarized according to thematic area.
Adherence to the Wakeful program | continuously for 9 weeks
  Adherence to the Wakeful program will be monitored and usage tracked continuously during the 9-week study. Data include the following:
  * Number of times a user: logs into the Wakeful app; opens the educational videos; opens the audio files; opens the audio files; acknowledges or comments on other users' reflections
  * Number of minutes a user spends: logged into the Wakeful app; on the educational videos; on the audio files; writing into the reflection text boxes; acknowledging or commenting on other users' reflections

SECONDARY OUTCOMES:
Change in mindful self-compassion | pre-intervention; post intervention
  Mindful self-compassion will be measured using the Self-Compassion Scale-12.
  This short form is a 12-item scale measuring items related to self-kindness, self-judgment, and common humanity. Statements on the Self-Compassion Scale are scored on a Likert scale of 1 (almost never) to 5(almost always). To calculate an overall compassion score - Items representing uncompassionate responses to inadequacy or suffering (the self-judgment, isolation, and over-identification subscales) are reverse-coded only when calculating the overall compassion score. In this way, higher scores represent a lower frequency of these responses.
Change in symptom burden of anxiety | pre-intervention; post intervention
  Symptom burden of anxiety will be measured at baseline and week 9 using the PROMIS 4-Item Short Forms of Anxiety. This 4-item scale measures uses a 5-point Likert scale (1=never to 5=always). The minimum value one can score is 4, and the maximum is 20. The lower scores represent better outcome.
Change in symptom burden of depression | pre-intervention; post intervention
  Symptom burden of anxiety will be measured at baseline and week 9 using the PROMIS 4-Item Short Forms of Depression. This 4-item scale measures uses a 5-point Likert scale (1=never to 5=always). The minimum value one can score is 4, and the maximum is 20. The lower scores represent better outcome.
Change in perceived stress | pre-intervention; post intervention
  Change in perceived stress will be measured using the Perceived Stress Scale-10.
  This short form is a 10-item scale measuring items related to perceived stress. Items are scored on a Likert scale of 0 (never) to 4(very often). Items representing unperceived stress responses are reverse-coded when calculating the overall score. In this way, lower scores indicate better outcome.
Change in health behaviors | pre-intervention; post intervention
  Change in health behaviors will be assessed using the Enacted Health Behaviors Questionnaire-10, a local questionnaire developed by the study researchers.
  Participants will report on the following: consumption frequency of red meat, grains, fruits and vegetables; use of cigarettes, tobacco products, and alcohol, preventive medications, vitamins, supplements, and medical screening tests; and engagement in regular physical exercise, meditation, and yoga. Unhealthy behaviors will be reverse scored. Higher scores represent better outcome. Significant change will be indicated by p<.05 on reported health behaviors between pre- and post-intervention.
Change in leisure time physical activity | pre-intervention; post intervention
  Change in leisure time physical activity will be measured using the Godin Leisure Time Exercise Questionnaire Physical Activity.
  This is a measure of self-reported physical activity participation. Participants report "times per week" they participate in strenuous (e.g., jogging), moderate (e.g., fast walking), and mild (e.g., easy walking) exercise over the past 7 days and the "average duration each time you exercised (in minutes)" for each of the three activity categories. Weekly minutes of total, light, moderate, and vigorous activity are calculated by multiplying the frequency and time of each activity. This value is divided by 7 to obtain daily averages. The minimum value one can score is 0, and the maximum depends on the number of self-reported minutes of physical activity. Higher scores indicate better outcome.

OTHER OUTCOMES:
Meditation experience in young adult cancer survivors | pre-intervention
  Meditation experience in young adult cancer survivors will be assessed using the Meditation Experience Questionnaire, a local questionnaire developed by the study researchers.
  Participants will report on their experience and familiarity with meditation concepts and practices. The measure uses Yes-No response options (1=Yes; 0=No). The minimum value one can score is 0, and the maximum is 5. The higher scores represent better outcome.
Treatment expectancy in young adult cancer survivors | pre-intervention
  Treatment expectancy in young adult cancer survivors will be assessed using the HEAL 6-Item Treatment Expectancy Subscale, a local questionnaire developed by the study researchers.
  Participants will report on the expectations they have about the outcomes of the study treatment. Each scale measure uses a 5-point Likert scale (1=not at all to 5=very much). The higher scores represent better outcome.
Socio-demographic and clinical factors in mindfulness program participation | pre-intervention
  Socio-demographic and clinical factors in mindfulness program participation in young adult cancer survivors will be assessed using the Socio-Demographic and Clinical Information Questionnaire., a local questionnaire developed by the study researchers.
  Participants will report on the following: age; sex; gender identity; relationship status; living status; education; employment; income; current/past health history; current/past cancer history and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: David E Victorson, PhD, Principal Investigator — Northwestern University; Siobhan M Phillips, PhD, MPH, Principal Investigator — Northwestern University
Locations (2):
- Northwestern University, Chicago, Illinois, United States
- Hospital Universitario San Ignacio Pontificia Universidad Jveriana, Bogotá, Capital District Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rabin C, Pinto B, Fava J. Randomized Trial of a Physical Activity and Meditation Intervention for Young Adult Cancer Survivors. J Adolesc Young Adult Oncol. 2016 Mar;5(1):41-7. doi: 10.1089/jayao.2015.0033. Epub 2015 Oct 15. PMID 26812450
- [Background] Meyer JD, Torres ER, Grabow ML, Zgierska AE, Teng HY, Coe CL, Barrett BP. Benefits of 8-wk Mindfulness-based Stress Reduction or Aerobic Training on Seasonal Declines in Physical Activity. Med Sci Sports Exerc. 2018 Sep;50(9):1850-1858. doi: 10.1249/MSS.0000000000001636. PMID 30113538
- [Background] Lucas AR, Focht BC, Cohn DE, Buckworth J, Klatt MD. A Mindfulness-Based Lifestyle Intervention for Obese, Inactive Endometrial Cancer Survivors: A Feasibility Study. Integr Cancer Ther. 2017 Sep;16(3):263-275. doi: 10.1177/1534735416668257. Epub 2016 Sep 14. PMID 27627985
- [Background] Ruffault A, Czernichow S, Hagger MS, Ferrand M, Erichot N, Carette C, Boujut E, Flahault C. The effects of mindfulness training on weight-loss and health-related behaviours in adults with overweight and obesity: A systematic review and meta-analysis. Obes Res Clin Pract. 2017 Sep-Oct;11(5 Suppl 1):90-111. doi: 10.1016/j.orcp.2016.09.002. Epub 2016 Sep 19. PMID 27658995
- [Background] Chatzisarantis NL, Hagger MS. Mindfulness and the intention-behavior relationship within the theory of planned behavior. Pers Soc Psychol Bull. 2007 May;33(5):663-76. doi: 10.1177/0146167206297401. Epub 2007 Apr 17. PMID 17440208
- [Background] Ulmer CS, Stetson BA, Salmon PG. Mindfulness and acceptance are associated with exercise maintenance in YMCA exercisers. Behav Res Ther. 2010 Aug;48(8):805-9. doi: 10.1016/j.brat.2010.04.009. Epub 2010 May 21. PMID 20488433
- [Background] Arch JJ, Craske MG. Mechanisms of mindfulness: emotion regulation following a focused breathing induction. Behav Res Ther. 2006 Dec;44(12):1849-58. doi: 10.1016/j.brat.2005.12.007. Epub 2006 Feb 7. PMID 16460668
- [Background] Kabat-Zinn J. An outpatient program in behavioral medicine for chronic pain patients based on the practice of mindfulness meditation: theoretical considerations and preliminary results. Gen Hosp Psychiatry. 1982 Apr;4(1):33-47. doi: 10.1016/0163-8343(82)90026-3. PMID 7042457
- [Background] Chambers R, Gullone E, Allen NB. Mindful emotion regulation: An integrative review. Clin Psychol Rev. 2009 Aug;29(6):560-72. doi: 10.1016/j.cpr.2009.06.005. Epub 2009 Jun 23. PMID 19632752
- [Background] Tsafou KE, De Ridder DT, van Ee R, Lacroix JP. Mindfulness and satisfaction in physical activity: A cross-sectional study in the Dutch population. J Health Psychol. 2016 Sep;21(9):1817-27. doi: 10.1177/1359105314567207. Epub 2015 Jan 28. PMID 25631662
- [Background] Sirois FM. A self-regulation resource model of self-compassion and health behavior intentions in emerging adults. Prev Med Rep. 2015 Mar 30;2:218-22. doi: 10.1016/j.pmedr.2015.03.006. eCollection 2015. PMID 26844074
- [Background] Mantzios M, Egan HH. On the Role of Self-compassion and Self-kindness in Weight Regulation and Health Behavior Change. Front Psychol. 2017 Feb 16;8:229. doi: 10.3389/fpsyg.2017.00229. eCollection 2017. No abstract available. PMID 28261147
- [Background] Schneider J, Malinowski P, Watson PM, Lattimore P. The role of mindfulness in physical activity: a systematic review. Obes Rev. 2019 Mar;20(3):448-463. doi: 10.1111/obr.12795. Epub 2018 Nov 23. PMID 30468299
- [Background] Hankin VV, Polster, R. Maximizing Acceptance and Enrollment in MBSR Randomized Controlled Trials with Older Men Diagnosed with Cancer. . Poster presented to the 8th Annual International Scientific Conference of Mindfulness in Medicine, Health Care, and Society Worcester, MA. 2010.
- [Background] Victorson D, Du H, Hankin V, et al. MINDFULNESS BASED STRESS REDUCTION DECREASES FEAR OF PROGRESSION OVER TIME FOR MEN WITH PROSTATE CANCER ON ACTIVE SURVEILLANCE: RESULTS FROM A RANDOMIZED CLINICAL TRIAL. The Journal of Urology. 2012;187(4S):384.
- [Background] Victorson D, Hankin V, Burns J, Weiland R, Maletich C, Sufrin N, Schuette S, Gutierrez B, Brendler C. Feasibility, acceptability and preliminary psychological benefits of mindfulness meditation training in a sample of men diagnosed with prostate cancer on active surveillance: results from a randomized controlled pilot trial. Psychooncology. 2017 Aug;26(8):1155-1163. doi: 10.1002/pon.4135. Epub 2016 May 3. PMID 27145355
- [Background] Victorson D, Maletich, C, Gutierrez, B, Schuette, S, Morgan, T, Kutikov, A, Kundu, S, Eggener, S, Brendler, C. Description of a New National Cancer Institute Funded Randomized Controlled Trial
- [Background] Victorson D. Redefining the psychosocial adjustment of young adults with cancer through mindfulness training: Results from a randomized controlled pilot trial. Psycho-Oncology. 2018;27:51.
- [Background] Maletich C CE, Gutierrez B, Schuette S, Sufrin N, Sanford S, Smith K, Victorson D. The effect of home practice on outcomes during an MBSR course for young adults with cancer: A mixed methods study. The Journal of Alternative and Complimentary Medicine. 2016;22(6):A83.
- [Background] Victorson D, Garland, E, Hanley, A, Greco, C. Is Mindfulness Immeasurable? Discovery and Dialogue of Conceptual, Practical, Scientific, and Experiential Solutions. Global Advances in Health and Medicine. 2018 7(1160):13.
- [Background] Victorson D, Maletich, C, Sufrin, N, Schuette, S, Gutierrez, B, Cordero, E, Johnson, C, Stencel, D, Bakosh, L, Ring, M. Development of a New Clinical Mindfulness Research Tool to Enhance, Deliver and Streamline Online Mindfulness Interventions. THE JOURNAL OF ALTERNATIVE AND COMPLEMENTARY MEDICINE. 2016;0(0):A21.
- [Background] Carmona-Fonseca J. [Demographic and epidemiologic changes in Colombia during the 20th century: facts and explanations]. Biomedica. 2005 Dec;25(4):464-80. Spanish. PMID 16433173
- [Background] Gaviria SL, Alarcon RD, Espinola M, Restrepo D, Lotero J, Berbesi DY, Sierra GM, Chaskel R, Espinel Z, Shultz JM. Socio-demographic patterns of posttraumatic stress disorder in Medellin, Colombia and the context of lifetime trauma exposure. Disaster Health. 2016 Nov 22;3(4):139-150. doi: 10.1080/21665044.2016.1263086. eCollection 2016. PMID 28265488
- [Background] Chaskel R, Gaviria SL, Espinel Z, Taborda E, Vanegas R, Shultz JM. Mental health in Colombia. BJPsych Int. 2015 Nov 1;12(4):95-97. doi: 10.1192/s2056474000000660. eCollection 2015 Nov. PMID 29093873
- [Background] Herran OF, Patino GA, Del Castillo SE. Dietary transition and excess weight in adults according to the Encuesta de la Situacion Nutricional en Colombia, 2010. Biomedica. 2016 Mar 3;36(1):109-20. doi: 10.7705/biomedica.v36i1.2579. PMID 27622444
- [Background] de Vries E, Buitrago G, Quitian H, Wiesner C, Castillo JS. Access to cancer care in Colombia, a middle-income country with universal health coverage. J Cancer Policy. 2018;15:104-112.
- [Background] Ferlay J, Colombet M, Soerjomataram I, Mathers C, Parkin DM, Pineros M, Znaor A, Bray F. Estimating the global cancer incidence and mortality in 2018: GLOBOCAN sources and methods. Int J Cancer. 2019 Apr 15;144(8):1941-1953. doi: 10.1002/ijc.31937. Epub 2018 Dec 6. PMID 30350310
- [Background] Mendieta CV, Gomez-Neva ME, Rivera-Amezquita LV, de Vries E, Arevalo-Reyez ML, Rodriguez-Ariza S, Castro E CJ, Faithfull S. Cancer as a Chronic Illness in Colombia: A Normative Consensus Approach to Improving Healthcare Services for those Living with and beyond Cancer and Its Treatment. Healthcare (Basel). 2021 Nov 29;9(12):1655. doi: 10.3390/healthcare9121655. PMID 34946381
- [Background] Victorson DK, M.; Maletich, C.; Lawton, R.C.; Hankin Kaufman, V.; Borrero, M.; Languido, L.; Lewett, K.; Pancoe, H.; Berkowitz, C. . A Systematic Review and Meta-Analysis of Mindfulness-Based Randomized Controlled Trials Relevant to Lifestyle Medicine. . American Journal of Lifestyle Medicine. 2015;9(3):185-211.
- [Background] Victorson D, Guitelman, J, DeArrudah, H, Van Hyfte, G, Pedersen, J, Oyola, S. Community-Engaged Yoga Research with Monolingual Spanish Speaking Women Diagnosed with Cancer: Findings from a Non-Randomized Pilot Study. Oral presentation at the 2017 Osher Integrative Medicine Research Conference. 2017;Chicago, IL.
- [Background] Banas JR, Victorson D, Gutierrez S, Cordero E, Guitleman J, Haas N. Developing a Peer-to-Peer mHealth Application to Connect Hispanic Cancer Patients. J Cancer Educ. 2017 Mar;32(1):158-165. doi: 10.1007/s13187-016-1066-6. PMID 27364905
- [Background] Victorson D, Banas J, Smith J, Languido L, Shen E, Gutierrez S, Cordero E, Flores L. eSalud: designing and implementing culturally competent ehealth research with latino patient populations. Am J Public Health. 2014 Dec;104(12):2259-65. doi: 10.2105/AJPH.2014.302187. Epub 2014 Oct 16. PMID 25320901